CLINICAL TRIAL: NCT01051115
Title: Dasatinib Combination for Chronic Lymphocytic Leukemia Patients With Chemo Refractory Disease
Brief Title: Dasatinib Combination for Chronic Lymphocytic Leukemia(CLL) With Refractory Disease
Acronym: D'ACCORD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, A.P. Kater, A.P. Kater, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D'Accord study
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; refractory; dasatinib; fludarabine
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasatinib (Experimental): Patients will be treated with dasatinib monotherapy 100mg daily. At four weeks patients will be re-evaluated. Patients with less than a partial response will receive fludarabine (orally 40mg/daily for 3 days q28) in addition to dasatinib.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Chemo-refractory CLL patients will be treated with dasatinib monotherapy 100mg daily.Patients with less than a partial response at 4 weeks will receive fludarabine (orally 40mg/daily for 3 days q28) in addition to dasatinib for a maximum of 6 cycles. Patients with at least a partial response will continue dasatinib monotherapy. Patients that receive monotherapy after the initial 28 days and that develop progressive disease will 'cross-over' to the combination treatment.
  Other Names: Sprycel; BMS-354825

SUMMARY:
Patients with chemo refractory CLL have a poor prognosis. 2 independent mechanisms are attributed to the development of chemoresistance in CLL. The first is a shift in the balance between pro- and anti-apoptotic regulators. The second mechanism is based on acquired mutations resulting in a dysfunctional p53 response. Recent studies indicate that the tyrosine kinase inhibitor dasatinib acts synergistically with both purine analogies and alkylating agents. Also, dasatinib has the potency to restore the apoptotic balance of CLL cells.

Hypothesis: Dasatinib will be clinically active in chemo-refractory CLL patients and will act synergistically with the purine-analogue fludarabine.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) is the most common leukemia in the western world. The disease mostly affects the elderly. At present no curative therapy is available. Although the majority of patients initially do respond to chemotherapy, most patients eventually develop drug resistance. The prognosis for patients with chemotherapy resistant disease is very poor wit an overall survival of approximately 10 months. Standard therapy for these patients currently does not exist. Treatment with the monoclonal antibody alemtuzumab could be tried, however toxicity of this drug is high especially following multiple cycles of chemotherapy. Allogeneic stem cell transplantation is still considered experimental in this setting and is only available for a minority of patients.

The development of chemoresistant disease is highly correlated with a disturbed balance of apoptosis regulating molecules, resulting in a decrease in sensitivity to apoptotic stimuli. The tyrosine kinase inhibitor dasatinib (Sprycel®) is successfully being used in the treatment of chronic myeloid leukemia (CML). This form of chronic leukemia is also characterized by a disturbed balance between apoptosis regulating genes, which can be restored by tyrosine kinase inhibitors. Recent studies indicate that also in CLL, dasatinib has the potential to restore the apoptotic balance. In this clinical study we will investigate whether dasatinib is an effective drug in the treatment of chemoresistant CLL and whether treatment with dasatinib restores the sensitivity to chemotherapeutic agents.

Objective of the study:

Primary:

To determine the response rate and response quality of dasatinib monotherapy or dasatinib/fludarabine combination in fludarabine refractory CLL patients

Secondary To asses the overall safety profile of this treatment approach To asses event free survival (i.e. time from registration to induction failure, progression, relapse or death whichever occurs first), progression free survival (i.e. time from registration to disease progression, relapse or death due to CLL whichever occurs first) and disease free survival (i.e. time from CR to relapse) To asses influence of dasatinib on the expression profile of apoptosis regulatory genes.

To determine whether dasatinib acts synergistically with other immuno-chemotherapeutic agents by co-culture experiments.

Study design:

Prospective, multi center clinical trial

Study population:

Patients with CLL in need of treatment AND fludarabine refractory, age 18-80 year inclusive

Intervention:

Patients will be treated with dasatinib monotherapy 100mg daily. At four weeks patients will be re-evaluated. Patients with less than a partial response will receive fludarabine (orally 40mg/daily for 3 days q28) in addition to dasatinib. After two cycles of fludarabine, responses will be evaluated. In case of progressive disease following 2 cycles of fludarabine in combination with dasatinib, patients will go off study. All other patients will be treated with four more cycles of fludarabine in combination with daily dasatinib treatment. Patients that receive monotherapy after the initial 28 days and that develop progressive disease will 'cross-over' to the combination treatment.

Primary study parameters/outcome of the study:

-- Clinical response rate and quality ( CR, PR) at 32 weeks

-In case of complete responses: minimal residual disease status

Secondary :

* Overall safety profile as determined by the incidence of clinically significant adverse events.
* Event free survival (i.e. time from registration to induction failure, progression, relapse or death whichever occurs first), progression free survival (i.e. time from registration to disease progression, relapse or death due to CLL whichever occurs first) and disease free survival (i.e. time from CR to relapse)

Extensive (functional) In vitro studies of dasatinib treated cells will be performed:

* Expression profile of apoptosis regulatory genes at the mRNA level (MLPA) and protein level (western blot)
* Study in vitro synergy of dasatinib treatment with different chemotherapeutic and immunotherapeutic drugs

Nature and extent of the burden and risks associated with participation, benefit and group relatedness (if applicable):

The monitoring of the patients during treatment and follow-up are according to the standard procedures in the treatment of patients with CLL. This means physical examination at a regular frequency (7 times from registration until the end of treatment; every 3 months during follow-up), blood sample analysis (9 times from registration until the end of treatment; every 3 months during follow-up), bone marrow analysis (2 times from registration until the end of treatment) and CT-scan (4 times from registration until the end of treatment). In addition, an ECG will be performed at entry of the study.

Hematological side-effects of dasatinib are cytopenias. Especially a drop in leukocytes and thrombocytes has been reported. In most cases, cytopenias can be controlled by dose adjustment. A temporarily inflammation of the liver can occur (< 3% of patients) and is in most cases reversible by dose adjustment. Most other reported side-effects are nausea, muscle cramps, painful joints, headache, fluid retention (including pleural effusion) and gain of weight. Most of the side-effects can successfully be managed by dose-adjustment.

Side-effects of fludarabine in the dose just in this study are temporarily cytopenias, nausea, emesis, diarrhea, mucositis, liver function abnormalities, fever, rash, conjunctivitis and dizziness.

ELIGIBILITY:
Inclusion Criteria:

* CLL confirmed according to the IWCLL Working Group criteria;
* Binet stages A or B with indication for treatment according to IWCLL guidelines, Binet C AND
* Fludarabine refractory, defined as relapse (any sign of disease recurrence or progression with or without indication for treatment ≤ 6 months following fludarabine containing chemo(immuno)therapy;
* Age 18-80 years inclusive;
* WHO performance status ≤ 2;
* No possibility for rapid reduced intensity allogeneic hematopoietic stem cell transplantation;
* At least 4 weeks without any treatment before study entry;
* Negative pregnancy test;
* Written informed consent;

Exclusion Criteria:

* Richter's transformation;
* Suspected or documented CNS involvement by CLL;
* Grade 3 cytopenia not due to bone marrow infiltration
* Concurrent medical condition which may increase the risk of toxicity, including:
* Pleural or pericardial effusion of any grade
* Cardiac Symptoms, including:
* Uncontrolled angina, congestive heart failure or MI within (6 months)
* Diagnosed congenital long QT syndrome
* Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
* prolonged QTc interval on pre-entry electrocardiogram (> 450 msec)
* Subjects with hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration;
* Severe pulmonary dysfunction (CTCAE grade III-IV);
* Active hepatitis B infection;
* History of significant bleeding disorder unrelated to the CLL, including:
* Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
* Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
* Ongoing or recent (within 3 months) significant gastrointestinal bleeding
* Known HIV positivity
* Clinically significant auto-immune hemolytic anemia (AIHA)
* Severe neurological or psychiatric disease;
* Significant hepatic dysfunction (Total bilirubin < 2.0 times ULN; Hepatic enzymes (AST, ALT ) ≤ 2.5 times ULN) except when caused by leukemic infiltration;
* Significant renal dysfunction (serum creatinine more than 150 uM/L after rehydration);
* History of active malignancy during the past 5 years with the exception of basal carcinoma of the skin or stage 0 cervical carcinoma;
* Concurrent use of CYP3A4 inducers or inhibitors, or QTc-prolonging agents*;
* Active, uncontrolled infections;
* Any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule;
* Female patients of reproductive potential who are not using effective contraception;
* The following medications should be considered for exclusion:

  1. Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Patients must discontinue drug 7 days prior to starting dasatinib) quinidine, procainamide, disopyramide amiodarone, sotalol, ibutilide, dofetilide erythromycin, clarithromycin chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, zyprasidone, cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.
  2. The concomitant use of H2 blockers or proton pump inhibitors with dasatinib is not recommended. The use of antacids should be considered in place of H2 blockers or proton pump inhibitors in patients receiving dasatinib therapy. If antacid therapy is needed, the antacid dose should be administered at least 2 hours prior to or 2 hours after the dose of dasatinib. Patient may not be receiving any prohibited CYP3A4

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2008-10; Primary Completion 2013-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
response rate and response quality | At 32 weeks of either dasatinib monotherapy or after 6 cycles of fludarabine and dasatinib combination

SECONDARY OUTCOMES:
overall safety profile of these treatment approaches, event free survival, progression free survival, relapse or death, disease free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Arnon P kater, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Marinus HJ van Oers, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (4):
- Netherlands (4):
  - Maastricht university medical center, Maastricht, Limburg
  - Academic Medical Center, Amsterdam, North Holland
  - University Medical Center Groningen, Groningen, Provincie Groningen
  - Erasmus MC-Daniel den Hoed Cancer Center, Rotterdam, South Holland

REFERENCES:
- See also: HOVON website — http://www.hovon.nl/working-groups/working-groups/chronical-lymfatic-leukemia.html